CLINICAL TRIAL: NCT03830424
Title: Assessment of Autonomic Nervous System Regulatory Mechanisms During Postnatal Period in Newborns
Brief Title: Assessment of Autonomic Nervous Regulation During Postnatal Period in Newborns
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Other Study IDs: EK69/2018
Record Dates: First submitted 2018-11-26; First posted 2019-02-05 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Infant, Newborn

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Healthy term newborns without pain relief during pain stimulus (intramuscular K vitamin administration and heel lancing for blood spot examination).
  Interventions: Procedure: Pain stimulus
- Sucrose group: Healthy term newborns with oral application of sucrose during pain stimulus (intramuscular K vitamin administration and heel lancing for blood spot examination).
  Interventions: Procedure: Pain stimulus; Dietary Supplement: Non-pharmacological pain relief
- Mother milk group: Healthy term newborns with oral application of mother milk during pain stimulus (intramuscular K vitamin administration and heel lancing for blood spot examination).
  Interventions: Procedure: Pain stimulus; Dietary Supplement: Non-pharmacological pain relief

INTERVENTIONS:
Procedure: Pain stimulus — Pain stimulus - intramuscular K vitamin administration, heel lancing = standard healthcare procedure
Dietary Supplement: Non-pharmacological pain relief — Administration of sucrose/mother milk during pain stimulus
  Groups: Mother milk group; Sucrose group

SUMMARY:
The project aims to assess the regulatory mechanisms of autonomic nervous system using noninvasive methods in newborns during postnatal adaptation period. Evaluated parameters will include complex analysis of electrodermal activity as a parameter reflecting sympathetic cholinergic system and indices of heart rate variability reflecting the activity of parasympathetic cardiac regulation. The project is focused on the neuro-psycho-physiological characteristics of physiological adaptation in early postnatal age and the effect of non-pharmacological pain relieving.

ELIGIBILITY:
Inclusion Criteria:

* healthy term newborns
* physiological postnatal adaptation
* signed parental informed consent

Exclusion Criteria:

* preterm delivery
* impaired postnatal adaptation
* perinatal infection
* congenital diseases and genetic anomalies
* hypoglycemia
* hyperbilirubinemia requiring phototherapy treatment

Ages: 1 Hour to 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy term newborns with physiological postnatal adaptation born in University Hospital in Martin (Slovakia).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Characteristics of parasympathetic (vagal) heart regulation in newborns in relation to nociception | within the first 4 days of postnatal life
  The study of cardiac vagal regulation of heart rate in relation to nociceptive stimulus using conventional linear and novel nonlinear analysis of heart rate variability (HRV) by special software (Kubios HRV, University of Eastern Finland, Kuopio, Finland). Continual recordings of RR intervals will be recorded using Polar V800 (Polar, Finland).
  HRV indices: linear (time domain - mean square of successive differences (MSSD); spectral domain - low frequency power (LF), high frequency power (HF), total spectral power (TP); non-linear (symbolic dynamics - 0V%, 2LV%, entropy).
Characteristics of sympathetic activity in newborns in relation to nociception | within the first 4 days of postnatal life
  The study of sympathetic cholinergic system indexed by electrodermal activity (EDA) using linear and novel nonlinear parameters characterizing complex sympathetic behavior in relation to nociceptive stimulus. Continual EDA recording associated with peripheral temperature monitoring will be performed using device BioInfinity, Thought Technology Ltd., Canada.
  EDA indices: linear - SCA (skin conductance amplitude), frequency of NS-EDR (nonspecific electrodermal responses), nonlinear - SIE (symbolic information entropy), and ApEn (approximate entropy).
Autonomic (parasympathetic) reactivity in response to non-pharmacological pain relief in newborns | within the first 4 days of postnatal life - during and after pain stimulus
  The study of autonomic nervous system complex regulatory mechanisms included in the reactivity - test: stress stimulus (painful intervention) with non-pharmacological pain relieving and recovery phase using HRV quantitative and qualitative analysis.
  1st group (control group, n=25) without pain relief; 2nd group (n=25) with oral application of sucrose during nociception stimulus; 3rd group (n=25) with oral application of mother milk during nociceptive stimulus.
Autonomic (sympathetic) reactivity in response to non-pharmacological pain relief in newborns | within the first 4 days of postnatal life - during and after pain stimulus
  The study of autonomic nervous system complex regulatory mechanisms included in the reactivity - test: stress stimulus (painful intervention) with non-pharmacological pain relieving and recovery phase using EDA quantitative and qualitative analysis.
  1st group (control group, n=25) without pain relief; 2nd group (n=25) with oral application of sucrose during nociception stimulus; 3rd group (n=25) with oral application of mother milk during nociceptive stimulus.
Pain quality assessment in newborns: Neonatal Facial Coding System (NFCS) scaling system | within the first 4 days of postnatal life - during pain stimulus
  Assessment of the pain quality during painful intervention in newborns associated with muscular application of K vitamin after birth and heel lancing (blood spot) on 3rd postnatal day (standard neonatal care) according to Neonatal Facial Coding System (NFCS).
  NFCS: visual monitoring of newborn's face during pain stimulus for the presence of 9 specific facial actions: brow bulge, eye squeeze, naso - labial furrow, open lips, stretch mouth (horizontal/vertical), lip purse, taut tongue, chin quiver.
  Scale range: 0 - 9 points; (0 = no pain; 9 = maximal pain presentation).

SECONDARY OUTCOMES:
Developmental aspect of parasympathetic regulatory mechanisms in early postnatal period | early after birth; 24 hours of life; 3rd - 4th day of life
  Assessment of the developmental aspect of cardiac vagal regulation indexed by HRV indices in relation to postnatal age (measures of HRV: early after birth; 24 hours of life; 3rd - 4th day of life).
Developmental aspect of sympathetic regulatory mechanisms in early postnatal period | early after birth; 24 hours of life; 3rd - 4th day of life
  Assessment of the developmental aspect of sympathetic cholinergic regulation indexed by EDA complex analysis in relation to postnatal age (early after birth; 24 hours of life; 3rd - 4th day of life).
Maternal clinical parameters effect on the neonatal autonomic (sympathetic) nervous system regulation | prior to delivery + retrospective data
  Study of the selected maternal clinical parameters [age (years), weight gain during pregnancy (kilograms), heart rate (beats per minute), systolic and diastolic blood pressure (millimeters of mercury) before delivery] in the interaction with sympathetic regulatory mechanisms - indexed by EDA.
Maternal clinical parameters effect on the neonatal autonomic (parasympathetic) nervous system regulation | prior to delivery + retrospective data
  Study of the selected maternal clinical parameters [age (years), weight gain during pregnancy (kilograms), heart rate (beats per minute), systolic and diastolic blood pressure (millimeters of mercury) before delivery] in the interaction with parasympathetic regulatory mechanisms - indexed by HRV.
Delivery mode effect on autonomic (sympathetic) nervous system regulation | at the time of delivery
  Study of the effect of delivery mode on the function and maturation of autonomic (sympathetic) nervous regulatory mechanisms - indexed by EDA.
Delivery mode effect on autonomic (parasympathetic) nervous system regulation | at the time of delivery
  Study of the effect of delivery mode on the function and maturation of autonomic (parasympathetic) nervous regulatory mechanisms - indexed by HRV.
Blood pressure in relation to autonomic (sympathetic) nervous system regulation | within the first 4 days of postnatal life
  Study of the relation between physiological parameters - blood pressure (systolic, mean, diastolic - in millimeters of mercury) and sympathetic regulatory mechanisms - indexed by EDA.
Blood pressure in relation to autonomic (parasympathetic) nervous system regulation | within the first 4 days of postnatal life
  Study of the relation between physiological parameters - blood pressure (systolic, mean, diastolic - in millimeters of mercury) and parasympathetic regulatory mechanisms - indexed by HRV.
Blood oxygen saturation in relation to autonomic (sympathetic) nervous system regulation | within the first 4 days of postnatal life
  Study of the relation between physiological parameters - blood oxygen saturation (in percentage) and sympathetic regulatory mechanisms - indexed by EDA.
Blood oxygen saturation in relation to autonomic (parasympathetic) nervous system regulation | within the first 4 days of postnatal life
  Study of the relation between physiological parameters - blood oxygen saturation (in percentage) and parasympathetic regulatory mechanisms - indexed by HRV.
Selected laboratory parameters in relation to autonomic (sympathetic) nervous system regulation | immediately after birth + on 3rd - 4th postnatal day
  Study of the effect of selected laboratory parameters [glycaemia (millimoles per liter), lactate (millimoles per liter), bilirubin (micromoles per liter)] on the sympathetic regulatory mechanisms - indexed by EDA.
Selected laboratory parameters in relation to autonomic (parasympathetic) nervous system regulation | immediately after birth + on 3rd - 4th postnatal day
  Study of the effect of selected laboratory parameters [glycaemia (millimoles per liter), lactate (millimoles per liter), bilirubin (micromoles per liter)] on the parasympathetic regulatory mechanisms - indexed by HRV.
Acid - base parameters in relation to autonomic (sympathetic) nervous system regulation | immediately after birth + on 3rd - 4th postnatal day
  Study of the effect of acid - base parameters [pH, pCO2 (kilopascals), base excess (millimoles per liler)] acquired immediately after birth on the sympathetic regulatory mechanisms - indexed by EDA.
Acid - base parameters in relation to autonomic (parasympathetic) nervous system regulation | immediately after birth + on 3rd - 4th postnatal day
  Study of the effect of acid - base parameters [pH, pCO2 (kilopascals), base excess (millimoles per liler)] acquired immediately after birth on the parasympathetic regulatory mechanisms - indexed by HRV.
Role of psychosocial factors in autonomic (sympathetic) nervous system regulation | immediately after birth + within the first 4 days of postnatal life
  Study of the effect of psychosocial factors (bonding, breastfeeding) on the sympathetic regulatory mechanisms - indexed by EDA.
Role of psychosocial factors in autonomic (parasympathetic) nervous system regulation | immediately after birth + within the first 4 days of postnatal life
  Study of the effect of psychosocial factors (bonding, breastfeeding) on the parasympathetic regulatory mechanisms - indexed by HRV.
Role of umbilical cord clamping in autonomic (sympathetic) nervous system regulation | at the time of delivery
  Study of the effect of immediate vs. delayed cord clamping on sympathetic regulatory mechanisms - indexed by EDA.
Role of umbilical cord clamping in autonomic (parasympathetic) nervous system regulation | at the time of delivery
  Study of the effect of immediate vs. delayed cord clamping on parasympathetic regulatory mechanisms - indexed by HRV.

CONTACTS AND LOCATIONS:
Overall Officials: Mirko Zibolen, Prof, MD, Study Director — Comenius University in Bratislava, Jessenius Faculty of Medicine in Martin
Locations (1):
- Jessenius Medical Faculty, Comenius University, Martin, Slovakia